CLINICAL TRIAL: NCT02062788
Title: Preoperative Oral Carbohydrate-rich Solution in Colorectal Cancer Patients: a Randomized Controlled Trial
Brief Title: Evaluation of Preoperative Oral Rehydration Solution in Colectomy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: patient enrollment was failed.
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Sung-Bum Kang, Associate Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORS-colectomy; B-1310/224-007 (Other: SNUBH IRB)
Record Dates: First submitted 2014-01-20; First posted 2014-02-14 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Insulin Resistance; Postoperative Complication
Keywords: Early Recovery After Surgery; Oral rehydration solution; Insulin resistance; Postoperative complication
MeSH Terms: conditions — Insulin Resistance; Postoperative Complications; Osteoarthritis | interventions — World Health Organization oral rehydration solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ORS group (Experimental): Oral rehydration solution (ORS) treated group
  Interventions: Dietary Supplement: Oral rehydration solution
- Non-ORS group (No Intervention): Oral rehydration solution (ORS) untreated group

INTERVENTIONS:
Dietary Supplement: Oral rehydration solution — Preoperative day #1: able to drink Oral rehydration solution (ORS) freely On day of Surgery: Allowed administration until 2hrs prior to surgery. 8AM patients(the first patients to undergo surgery of the day) are recommended to administer ORS at 5:30AM
  Other Names: NoNPO (Daesang)
  Arms: ORS group

SUMMARY:
Elective colectomy procedures typically require bowel preparation starting 2 days prior to the surgery. Osmotic laxatives such as Colyte® are administered 2 days prior, and Nothing by mouth (NPO) is required 1 day prior to ensure no fecal residue is left in the bowel. Though it may ensure a cleaner and safer surgery, this longer period of starvation increases insulin resistance and may increase post-op complications. However, there is evidence that administration of oral rehydration solution(ORS) prior to surgery reduces insulin resistance. Our purpose is to evaluate the difference of insulin resistance in those who received ORS 1 day prior to surgery and those who did not.

DETAILED DESCRIPTION:
1. Enhanced Recovery After Surgery (ERAS) Enhanced Recovery After Surgery(ERAS) was introduced in the early 2000s by Kehlet et.al., and was applied primarily to patients receiving colectomy. As the knowledge and understanding of this concept continues to grow, we are now able to change the way we treat pre- and post- operative patients. In Europe, it has been proven that applying this concept to patients resulted in decreased length of post-operative hospital stay, post-op complications and overall hospital costs.
2. The change in HOMA-IR with shorter preoperative Nothing by mouth (NPO) period in ERAS patients

   1. HOMA-IR Index equation (evaluation of Insulin resistance)

      = Insulin (μU/ml) X blood glucose (mg/dl) / 405
   2. HOMA-IR was statistically proven to have been lowered in patients who received ORS 2hr prior to surgery.
   3. Reference

      * Increased insulin resistance induces hyperglycemia
      * Toxicity of post-op hyperglycemia and their relation to post-op complications
      * Insulin resistance increases in procedures such as herniorrhaphy or laparoscopic cholecystectomy. Administration of preoperative carbohydrates decrease post-op nausea and vomiting
      * Conventional pre-op 8hr fasting increases insulin resistance and influences increased glucose levels
3. Additional benefits of shorter preoperative fasting

   1. Relieve of stress of fasting
   2. Help stabilize post-op triglyceride, cortisol, and glucose levels
   3. Reduce infectious complications

ELIGIBILITY:
Inclusion Criteria:

* ASA grade I~II (DM, CVA, COPD, ESRD, MI, TIA etc. excluded)
* Age: adults age 19~75
* Patients undergoing elective colon cancer surgery
* Able to take the ORS per orally. Able to swallow without trouble of aspiration tendencies
* BMI of less than 27.5
* Child-Turcotte-Pugh Classification score of less than 6

Exclusion Criteria:

* emergency cases such as obstruction or perforation
* food allergy
* abdominal distension at present
* prior gastric surgery

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-02; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Changes in HOMA-IR levels | 6hr, 24hr, 48hr
  HOMA-IR = Insulin (μU/ml) X blood glucose (mg/dl) / 405 insulin and glucose levels are obtained 6hrs, 24hrs, 48hrs post-op Derive the value using the obtained sample variables into the HOMA-IR equation and comparison using statistical analytic methods

SECONDARY OUTCOMES:
Changes in Insulin levels | 0hr (induction of general anaesthesia), postop 6hr, 24hr, 48hr
Changes in glucose level | 0hr (induction of general anaesthesia), postop 6hr, 24hr, 48hr
Changes in cortisol level | 0hr (induction of general anaesthesia), postop 6hr, 24hr, 48hr
Assessment of patient pain via Visual Analogue Scale | Participants will be evaluated daily till discharge, an expected average of 6 days
Reduction of postoperative complications | Participants will be evaluated daily till discharge, an expected average of 6 days
Changes in triglyceride level | 0hr (induction of general anesthesia), 24hr

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Bum Kang, Ph.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea